CLINICAL TRIAL: NCT03764306
Title: New Ischemic Cerebral Lesions Revealed by the Imaging Magnetic Resonance Imaging After Endarterectomy vs. Stenting Under Proximal Protection for the Treatment of Symptomatic Carotid Stenosis: Results of a Randomised Prospective Trial
Brief Title: New Ischemic Cerebral Lesions After Endarterectomy vs. Stenting for the Treatment of Symptomatic Carotid Stenosis
Acronym: CARECarotid
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problem with recruitment of patients meeting the inclusion criteria.
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Pawel Latacz, Principal Investigator, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 137/KBL/OIL/2015
Record Dates: First submitted 2018-11-29; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Carotid Artery Stenosis; Carotid Atherosclerosis; Stroke, Ischemic
Keywords: carotid angioplaty; MRI DWI
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases; Ischemic Stroke | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to one of the two treatment arms: surgical endarterectomy or carotid angioplasty with stenting under proximal protection
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carotid Artery Stenting (Active Comparator): Subjects will undergo carotid artery angioplasty and stenting with any CE-certificated carotid stent with a proximal protection system Mo.Ma
  Interventions: Procedure: Carotid Artery Stenting
- Endarterectomy carotid artery (Active Comparator): Subjects will undergo carotid endarterectomy
  Interventions: Procedure: Endarterectomy carotid artery

INTERVENTIONS:
Procedure: Carotid Artery Stenting — Carotid artery stenting was considered successful if there was no residual stenosis greater than 20%, and there was no dissection of target artery following the procedure.
  Arms: Carotid Artery Stenting
Procedure: Endarterectomy carotid artery — Surgical endarterectomy was considered successful if there was no residual stenosis after procedure, without symptoms.
  Arms: Endarterectomy carotid artery

SUMMARY:
Background and purpose. Even if periprocedural cerebral microembolism associated with carotid endarterectomy or stenting usually does not manifest as clinically overt stroke, neuropsychological disturbances resulting from these events represent an important clinical and socioeconomic problem. Still, it remains unclear whether the use proximal protection can lower the incidence of cerebral embolism associated with the treatment of carotid stenosis.

Materials and methods. This was a prospective randomised single-centre study, which was aimed at comparison of surgical eversion endarterectomy with stenting under proximal protection in symptomatic patients. The investigators evaluated the incidence of new ischaemic lesions revealed by the diffusion-weighted magnetic resonance imaging 2-4 days after the treatment and neurologic events.

DETAILED DESCRIPTION:
The CARECarotid was a prospective randomised single-centre study, which was performed in the University Hospital in Kraków. It was planned to evaluate 50 patients presenting with symptomatic lesions of the internal carotid artery.

Patients were randomly assigned to one of the two treatment arms: surgical endarterectomy or carotid angioplasty with stenting under proximal protection. All patients provided their written informed consent to undergo the procedures and to participate in this trial.

In all surgical patients carotid endarterectomy will perform using the eversion technique. All surgical endarterectomies will perform under cervical block anaesthesia.

Perioperatively patients in the surgical arm received aspirin; other antiplatelet or anticoagulant agents were not administered during 5 days before surgery.

All procedures in carotid artery stenting will perform with proximal protection system - the Mo.Ma (Medtronic, Minneapolis, MN, USA) device. The investigators will implante stents that were tailored to the localisation of lesions and morphology of carotid arteries: Carotid Wallstent (Boston Scientific, Natick, MA, USA, and in patients with tortuous arteries Precise Pro RX (Cordis, Fremont, CA, USA) or Roadsaver (Terumo, Tokyo, Japan). Patients in the stent arm will receive clopidogrel 75 mg/day and aspirin 75 mg/day. These drugs were administered during 3 days before planned procedure and then 3-6 months after stent implantation. All patients will have MRI DWI performed before and 2-4 days after procedures in both groups. Within 6 months there will be an evaluation of the incidence of neurological events.

ELIGIBILITY:
Inclusion criteria comprised:

* patient's age ≥ 18 years;
* 60-99% stenosis of the internal carotid artery (degree of stenosis assessed by means of Doppler sonography, CT angiography or catheter angiography);
* diameter of the target internal carotid artery not more than 7 mm;
* symptomatic lesion (a history of ipsilateral stroke, transient ischaemic attack or reversible ischaemic neurological deficit);
* localisation and morphology of the lesion making possible surgical eversion endarterectomy or endovascular angioplasty with stent implantation;
* written informed consent.

Exclusion criteria comprised:

* target lesion that has been previously stented;
* highly calcified lesions;
* very tortuous common and internal carotid arteries;
* occlusion of the contralateral carotid artery without adequate collateral circulation through the circle of Willis (revealed by means of transcranial Doppler sonography);
* anatomical contraindications for eversion endarterectomy;
* acute ipsilateral stroke;
* disabling stroke at any side;
* other severe pathologies of the brain resulting is significant loss of cerebral tissue and/or significant neurological deficits, such as extensive previous stroke or multiple lacunar infarcts;
* history of haemorrhagic transformation of ischaemic stroke;
* severe comorbidities (such as cancer or decompensated heart failure);
* allergy to aspirin, clopidogrel or ticlopidine;
* allergy to iodinated contrast media;
* pregnant women;
* women of reproductive age who do not use effective contraception;
* metallic implants (such as peacemakers and orthopaedic endoprostheses) or other known contraindications for magnetic resonance imaging;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is to compare the rate of new ischemic brain injury detectable on MRI after carotid artery stenting and endarterectomy. | 2-4 days after procedure
  Number of patients with treatment related new ipsilateral cerebral embolic lesions in brain diffusion-weighted magnetic resonance imaging within 2-4 days post carotid artery stenting and endarterectomy. Number, size and location new cerebral lesions per patients in both groups.

SECONDARY OUTCOMES:
Any Stroke, TIA, MI or death | 6 months
  Number of patients with occurrence of any stroke, transient ischemic attack (TIA), myocardial infarction, or death within 6 months after carotid artery stenting and endarterectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Latacz, PhD MD, Principal Investigator — Jagiellonian University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cremonesi A, Gieowarsingh S, Spagnolo B, Manetti R, Liso A, Furgieri A, Barattoni MC, Ghetti L, Tavazzi L, Castriota F. Safety, efficacy and long-term durability of endovascular therapy for carotid artery disease: the tailored-Carotid Artery Stenting Experience of a single high-volume centre (tailored-CASE Registry). EuroIntervention. 2009 Nov;5(5):589-98. doi: 10.4244/eijv5i5a95. PMID 20142180
- [Result] Ansel GM, Hopkins LN, Jaff MR, Rubino P, Bacharach JM, Scheinert D, Myla S, Das T, Cremonesi A; Investigators for the ARMOUR Pivotal Trial. Safety and effectiveness of the INVATEC MO.MA proximal cerebral protection device during carotid artery stenting: results from the ARMOUR pivotal trial. Catheter Cardiovasc Interv. 2010 Jul 1;76(1):1-8. doi: 10.1002/ccd.22439. PMID 20222019
- [Result] Bersin RM, Stabile E, Ansel GM, Clair DG, Cremonesi A, Hopkins LN, Nikas D, Reimers B, Sievert H, Rubino P. A meta-analysis of proximal occlusion device outcomes in carotid artery stenting. Catheter Cardiovasc Interv. 2012 Dec 1;80(7):1072-8. doi: 10.1002/ccd.24433. Epub 2012 Jul 23. PMID 22454248
- [Result] Gao MY, Sillesen HH, Lorentzen JE, Schroeder TV. Eversion carotid endarterectomy generates fewer microemboli than standard carotid endarterectomy. Eur J Vasc Endovasc Surg. 2000 Aug;20(2):153-7. doi: 10.1053/ejvs.1999.1072. PMID 10942686
- [Result] Silver FL, Mackey A, Clark WM, Brooks W, Timaran CH, Chiu D, Goldstein LB, Meschia JF, Ferguson RD, Moore WS, Howard G, Brott TG; CREST Investigators. Safety of stenting and endarterectomy by symptomatic status in the Carotid Revascularization Endarterectomy Versus Stenting Trial (CREST). Stroke. 2011 Mar;42(3):675-80. doi: 10.1161/STROKEAHA.110.610212. Epub 2011 Feb 9. PMID 21307169